CLINICAL TRIAL: NCT04208490
Title: Implementation and Effectiveness Trial of HN-STAR
Acronym: HN-STAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00060694; NCI-2019-03600 (Registry Identifier: NCI CTRP); WF-1805CD (Other: WF NCORP RB); 5UG1CA189824 (NIH)
Record Dates: First submitted 2019-12-04; First posted 2019-12-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: Survivorship
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HN-STAR (Other)
  Interventions: Other: HN-STAR Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Other: HN-STAR Intervention — The Head and Neck Survivorship Tool (HN-STAR) is a web-based tool used to assist clinicians in implementing the ACS/ASCO HNC survivorship guidelines.
  Arms: HN-STAR

SUMMARY:
People who have been treated for head and neck cancer (HNC survivors) can experience serious consequences from their cancer and its treatment, ongoing risks of new cancers, and other unrelated illnesses. These concerns pose challenges to the provision of comprehensive care to HNC survivors. We created HN-STAR to facilitate and tailor the ongoing care of HNC survivors. Survivors use HN-STAR on a computer or tablet to answer questions about symptoms and health concerns before a routine visit with a cancer care provider. During the clinic visit, the provider uses HN-STAR to see evidence-based recommendations for managing each concern reported by the survivor. The provider and survivor discuss recommendations and select appropriate actions (e.g., testing, referrals, prescriptions, self-management). HN-STAR produces a survivorship care plan that includes all reported concerns and the actions selected in clinic. The survivorship care plan is given to the survivor and the primary care provider. Three months, six months, and nine months later, the survivor uses HN-STAR from home (or clinic) to report their concerns again, and a new survivorship care plan is created each time.

Our trial randomizes 20-36 oncology practices from the National Community Oncology Research Program to use HN-STAR or provide usual care to 298-400 recent survivors of head and neck cancer. We hypothesize that survivors in the HN-STAR arm will have greater improvement in patient-centered outcomes (including cancer-related well-being, symptoms, and patient activation) over one year compared to survivors in the usual care arm, measured by surveys at baseline and one year later. We also hypothesize that survivors in the HN-STAR arm will be more likely to receive care that is aligned with evidence-based recommendations during the year of the study than survivors in the usual care arm. Our final aim investigates the implementation of HN-STAR in clinical practice, using interviews and surveys of survivors, providers, and other clinic staff to understand the feasibility, acceptability, appropriateness, and other aspects of providing survivorship care to head and neck cancer survivors.

ELIGIBILITY:
Survivor Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of primary or locoregionally recurrent head and neck squamous cell carcinoma, specifically oral cavity, larynx, oropharynx, hypopharynx, and unknown squamous cell carcinoma primary.
* Completed chemotherapy and/or radiation therapy with curative intent for head and neck squamous cell carcinoma ≤ 24 months prior to designated clinician visit.
* Deemed free of disease at last assessment.
* Cognitively and physically able to complete study survey per local NCORP site staff discretion.
* Scheduled for a clinic visit with a provider who has agreed to participate in this study and meets requirements for the arm to which their practice has been assigned (the practice designated clinician) for routine follow-up.
* Willing to complete study assessments 3, 6, and 9 months after the designated clinic visit either 1) remotely (via telephone or videoconference using smartphone, tablet, or computer) or 2) at the clinic to complete study assessments on a clinic tablet or computer.

Survivor Exclusion Criteria:

* In active cancer treatment (including hormone therapy) for any other cancer, excluding local therapy for non-melanoma skin cancer.
* Evidence of prior cancer (excluding non-melanoma skin cancer) within 3 years of the designated clinician visit.
* Head and neck tumor histology of lymphoma, adenocarcinoma or melanoma.
* Recurrent, persistent, or progressive disease at last assessment (per scan or clinical assessment).
* Does not speak or read English, because the HN-STAR tool is only available in English at this time.
* Received only surgery as treatment for head and neck cancer.
* Current, planned enrollment, or in follow-up on another interventional symptom management study protocol, as per patient self-report or research staff members' knowledge at the time of consent. Concurrent participation in treatment or imaging studies is allowed.

Designated Clinician Inclusion Criteria:

* Age > = 18 years
* MD, DO, NP, or PA
* Able to speak and read English, because the HN-STAR tool is only available in English at this time.
* Routinely provides care for cancer patients or survivors.
* Willing to complete study-specific trainings and incorporate HN-STAR or provide usual care in a routine follow-up care visit

Stakeholders Inclusion Criteria:

* Age > = 18
* Member of the practice clinical or administrative team who is involved in the oversight of the delivery of head and neck cancer survivorship care or who would make decisions about implementing head and neck survivorship tools such as HN-STAR. This could include clinic administrators, nurse navigators, key clinical team members, program directors, and other staff (e.g., service line or nursing leaders).
* Employed for at least one month at the practice.
* Able to speak and reads English, because the HN-STAR tool is only available in English at this time.

Stakeholder Exclusion Criteria:

* Is the designated clinician at the practice.

Primary Care Provider Inclusion Criteria:

* Provides primary care (general preventative care) to a survivor enrolled in the HN-STAR study.
* Age >= 18
* MD, DO, NP, or PA

Primary Care Provider Exclusion Criteria:

* Provides Oncology Care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HNC-Specific QOL | Baseline & 1 year
  Measured using Trial Outcome Index from the Functional Assessment of Cancer Therapy Head and Neck. It is a 23-item summary measure that ranges from 0 to a maximum of 96 where higher scores indicate better overall physical and functional outcomes.

SECONDARY OUTCOMES:
Change in QoL | Baseline & 1 year
  Measured using domains and overall measures from the FACT H&N. The total score evaluates overall QoL in Head and Neck Cancer patients and ranges from 0 to 144, with higher scores indicating better overall QoL. Subscales are calculated by summing the relevant questions [answered using a Likert scale ranging from 0 (Not at all) to 4 (Very much)]. Higher scores on subscales represent a better health state.
Change in QoL | Baseline & 1 year
  Measured using scales from the EORTC QLQ-C30. Scales from the EORTC QLQ-C30 evaluate functional status, global health status and symptoms. All scales range from 0 to 100, with higher scores representing higher functioning, QoL or symptoms.
Change symptom burden | Baseline & 1 year
  Measured using scales from the EORTC QLQ-HN43. Symptom subscales from the EORTC QLQ- HN43 range from 0 to 100, with higher scores representing higher symptom burden.
Change in symptom burden | Baseline & 1 year
  Measured using PRO-CTCAE items for relevant symptoms.
Change in pain | Baseline & 1 year
  Measured using Brief Pain Inventory Short Form. Pain severity and interference items are measured using a scale from 0 to 10, with higher scores indicating worse pain or interference. The average is used as a summary measure of pain severity and pain interference.
Change in patient activation | Baseline & 1 year
  Measured using Patient Activation Measure Short Form. PAM score ranges from 0 to 100, with higher score meaning higher level of activation.
Change in perceived quality of cancer care | Baseline & 1 year
  Measured using the CAHPS® Cancer Care Survey.
Adherence and surveillance of guideline concordant care | These variables will be derived from the medical record during the year following the initial visit.
  Rate at which survivors had ≥1 visit to a primary care provider in the year following the initial visit will be compared by arm. Receipt or non-receipt of guideline-concordant cancer surveillance will be derived from the oncology medical records and compared by arm.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - John H Stroger Jr Hospital Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Reid Health, Richmond, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Maine Medical Partners Otolaryngology, Portland, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Licking Memorial Hospital, Newark, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Aspirus Langlade Hospital, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu
URL: https://nctn-data-archive.nci.nih.gov/